CLINICAL TRIAL: NCT00367770
Title: A Multi-Center, Open-Label Extension Study to Protocol AC-052-405 to Evaluate the Safety and Efficacy of Tracleer (Bosentan) in Patients With Pulmonary Arterial Hypertension Related to Eisenmenger Physiology
Brief Title: BREATHE 5-OL: Tracleer (Bosentan) in Patients With Pulmonary Arterial Hypertension Related to Eisenmenger Physiology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-409
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: bosentan; PAH related to Eisenmenger physiology; Tracleer
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tracleer (Experimental): The starting dose for all patients will be 62.5 mg b.i.d. At the Week 4 visit, patients who were started on 62.5 mg b.i.d. will be uptitrated to 125 mg b.i.d. if the 62.5 mg b.i.d. dose was well-tolerated.
  Interventions: Drug: Tracleer®

INTERVENTIONS:
Drug: Tracleer® — Patients will receive up to 125 mg b.i.d. of Tracleer.

SUMMARY:
This 6-month open label study will evaluate the long term safety of bosentan (via oxygen saturation) and efficacy (exercise capacity) in patients who have completed the BREATHE-5 study (PAH related to Eisenmenger physiology). Treatment duration is 6 months.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single -arm study with bosentan, initial dose of 62.5 mg b.i.d., with a target dose of 125 mg b.i.d. All patients will be assessed for eligibility during the baseline visit (same as Week 16, end of study BREATHE-5 visit), and will have the option to enter into the open-label extension study at a starting dose of 62.5 mg b.i.d., for safety reasons. Visit 2 is required as a safety visit to assess oxygen saturation (SpO2) after 1 week of bosentan treatment. Patients will return for Visit 4 after 4 weeks of treatment, and the dose will be up-titrated to 125 mg b.i.d. or maintained at 62.5 mg b.i.d. at the judgement of the investigator. Data will be collected for a total of 24 weeks or until the sponsor decides to stop the study. If the results from Study AC-052-403 or AC-052-405 demonstrate significant safety issues, this extension study may be terminated at the sponsor's request.

ELIGIBILITY:
Inclusion Criteria:

1. Patients stable with PAH upon completion of the BREATHE-5 randomized, double-blind, placebo- controlled 16-week study.
2. For female patients, only non-pregnant women who are surgically sterile, postmenopausal or have documented infertility (over 50 years of age and amenorrheic for at least 1 year), or those of childbearing potential using one of the following methods of contraception: Barrier-type devices (e.g., condom, diaphragm) used ONLY in combination with a spermicide. A double-barrier method is recommended; intrauterine devices (IUDs); oral or implanted contraceptives, if used in combination with a barrier method.
3. Patients providing written informed consent.

Exclusion Criteria:

1. Patients who withdrew prematurely from BREATHE-5, AC-052-405.
2. Patients who are pregnant or nursing.
3. Patients who are receiving epoprostenol or prostacyclin analogues, or are expected to receive any of these drugs during the study.
4. Patients with AST and/or ALT values greater than 3 times the upper limit of normal.
5. Patients with hemoglobin or hematocrit that is more than 30% below the normal range (patients with secondary polycythemia are permitted in the study).
6. Patients with systolic blood pressure < 85 mm Hg.
7. Patients taking phosphodiesterase inhibitors, other endothelin receptor antagonists or are receiving another investigational product.
8. Patients active on organ transplant list.
9. Patients who are receiving or expected to receive glyburide, cyclosporin A or tacrolimus.
10. Patients not able to comply with the protocol or adhere to therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Landzberg, MD, Study Chair — BACH Pulmonary Hypertension Service, Boston, U.S.A.
Locations (17):
- United States (2):
  - BACH Pulmonary Hypertension Service, Boston, Massachusetts
  - Texas Children's Hospital, Houston, Texas
- Australia (2):
  - Royal Prince Alfred Hospital - Central Clinical School, Camperdown
  - The Royal Melbourne Hospital, Victoria
- Universitatsklinikum fur Innere Medizin II, Vienna, Austria
- UZ Gasthuisberg, Leuven, Belgium
- Canada (2):
  - The Peter Lougheed Centre, Calgary, Alberta
  - Toronto General Hospital, Toronto, Ontario
- Hospital Necker-Enfants Malades, Paris, France
- Germany (2):
  - Herzzentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum Munchen, München
- Italy (2):
  - University of Bologna, Bologna
  - San Matteo Hospital, Pavia
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Unidad Medico Quirurgica de Cardiologia - Edificio General, Madrid, Spain
- United Kingdom (2):
  - Scottish Vascular Unit - Western Infirmary, Glasgow
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight centers in six countries: Germany (1), Italy (2), the Netherlands (1), Spain (1), U.K. (2), U.S.A. (1)
  Patients with stable PAH upon completion of the BREATHE-5 randomized, double-blind, placebocontrolled 16-week study were given option to enter into the open-label extension study.
Period: Overall Study
Arm/Group | Tracleer
Started | 37
Completed | 35
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walk Distance
Time Frame: from baseline to week 24
Population: The analysis was done in the safety set.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 35
m | 13.5 (57.2)

2. Primary Outcome: Change in Borg Dyspnea Index
Description: Borg scale a numerical scale for assessing dyspnea, from 0 representing no dyspnea to 10 as maximal dyspnea.
Time Frame: from baseline to week 24
Population: The analysis was done in the safety set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 35
units on a scale | 0.1 (1.4)

3. Primary Outcome: Number of Participants With a Change in WHO Functional Class
Description: Number of participants with a change in WHO functional class from baseline to week 24.
  A change from a higher to a lower functional class (i.e. III to II, III to I or II to I) is considered as an improvement.
Time Frame: from baseline to week 24
Population: The analysis was done in the safety set.
Measure: Number; unit: participants
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 35
participants | 13

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Tracleer
Serious Adverse Events (participants affected / at risk) | 7/37
Other Adverse Events (participants affected / at risk) | 25/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tracleer (N=37)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1
LETHARGY (Nervous system disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
sudden death (General disorders) | 1
rectal hemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tracleer (N=37)
OEDEMA PERIPHERAL (General disorders) | 7
CHEST PAIN (General disorders) | 4
FATIGUE (General disorders) | 2
NASOPHARYNGITIS (Infections and infestations) | 5
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
VIRAL INFECTION (Infections and infestations) | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2
PALPITATIONS (Cardiac disorders) | 2
DIZZINESS (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 2
DIARRHOEA (Gastrointestinal disorders) | 3
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2
GOUT (Metabolism and nutrition disorders) | 2
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less